CLINICAL TRIAL: NCT06923371
Title: Investments in Mothers' and Babies' Health and Well-being During Pregnancy, Perinatal and Post-natal Period: Evidence From an Unconditional Cash Allowance Program in the Appalachian Region, USA, 2024-2027
Brief Title: Moms and Babies Health and Well-being
Acronym: MBHW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: The Bridge Project (Unknown)
Responsible Party: Principal Investigator, Catherine Monk, Chief, Division of Women's Mental Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAV2019; BP CU24-1156 (Other Grant/Funding Number: The Bridge Project)
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Maternal and Child Health Outcomes
Keywords: unconditional cash transfers; maternal health; child health; pregnancy outcomes; postpartum health; healthcare access; nutrition; social determinants of health; cash allowance program; perinatal health
MeSH Terms: interventions — Infant Health

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The Columbia research team will be blinded to intervention status excluding the PI and the Data Manager.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fee group (Other): Participants in the high-fee group will receive a larger monetary allowance to evaluate the impact of increased financial support on the health outcomes of pregnant women and their babies. This intervention will assess whether greater financial resources during pregnancy and early infancy improve baby growth, maternal well-being, healthcare access, and healthier decision-making.
  Interventions: Behavioral: Direct Cash Support for Maternal and Infant Health (High fee)
- Low fee group (Other): Participants in the low-fee group will receive a smaller monetary allowance to explore the impact of moderate financial support on maternal and infant health outcomes. The intervention will assess whether financial assistance during pregnancy and early infancy improves baby growth, maternal well-being, healthcare access, and healthier food choices. By comparing this group to the high-fee group, the researchers aim to understand how different levels of financial support affect health outcomes in economically challenged populations.
  Interventions: Behavioral: Behavioral: Direct Cash Support for Maternal and Infant Health (Low fee)

INTERVENTIONS:
Behavioral: Direct Cash Support for Maternal and Infant Health (High fee) — The high fee group will receive direct cash assistance to pregnant women and mothers of infants to improve access to healthcare, alleviate financial strain, and facilitate healthier lifestyle choices. This group will receive a higher level of financial support compared to the low fee group, with the aim of examining how larger amounts of financial assistance affect maternal and infant health, healthcare access, and well-being.
  Arms: High fee group
Behavioral: Behavioral: Direct Cash Support for Maternal and Infant Health (Low fee) — The low fee group will receive direct cash assistance to pregnant women and mothers of infants to improve access to healthcare, reduce financial strain, and support healthier lifestyle choices. This group will receive a lower level of financial support compared to the high fee group, allowing us to compare the effects of varying levels of financial assistance on maternal and infant health outcomes.
  Arms: Low fee group

SUMMARY:
The goal of this clinical trial is to see how giving direct cash support affects the health of pregnant women and their babies in the U.S. Many families, especially those with low incomes, face challenges during pregnancy and after childbirth. This study will explore whether financial help during these times leads to better health.

The main questions this research aims to answer are:

* Does extra money during pregnancy and a baby's first months improve the baby's growth and overall health?
* How does financial support affect a mother's physical and mental health before and after birth?
* Does having extra money help moms get better healthcare and make healthier food choices for themselves and their babies?

Participants in this study will be randomly assigned to either a high cash or low cash group. They will be enrolled in the study and asked to complete:

* A baseline survey
* A follow-up survey 12 months after enrollment
* A final survey 18 months after enrollment

In addition, participants' medical records will be reviewed, and some may be selected for a qualitative interview to share more about their experiences.

This research is being done in partnership with The Bridge Project, a program that helps moms in need. The goal is to find better ways to support the health of moms and babies facing financial hardship.

DETAILED DESCRIPTION:
In 2022, the United States witnessed a concerning statistic: approximately 1 in 5 children lived in poverty, marking the highest child poverty rate among high-income countries. This figure becomes even more alarming when examining specific demographic groups. Research from the Center on Budget and Policy Priorities reveals that 1 in 2 Black and Latino households with children reported financial hardships, compared to 1 in 4 white households with children. Furthermore, Black children were nearly three times as likely to live in poverty as White children in 2017, even after accounting for government assistance. According to the Census Bureau, the expiration of pandemic-related social support programs at the end of COVID-19 coincided with a dramatic increase in the national child poverty rate, which surged from 5.2% in 2021 to 12.4% in 2022.

Simultaneously, maternal mortality, particularly among impoverished pregnant women, has become a pressing public health issue. Over the last three decades, the maternal mortality rate in the U.S. has doubled from 7 per 100,000 live births in 1986 to 17 per 100,000 in 2016, with disproportionately higher rates among Black and Brown women. During the COVID-19 pandemic, the National Center for Health Statistics reported an 18.4% increase in deaths during pregnancy or the post-natal period in 2019 and 2020. According to the Centers for Disease Control and Prevention (CDC), 4 in 5 of these deaths were preventable, with the leading causes being mental health conditions (23%), hemorrhage (14%), cardiac and coronary conditions (13%), and infections (9%). Studies have emphasized the critical role of social determinants of health, such as access to care, food security, housing, and safety, in influencing maternal mortality outcomes. Addressing these factors is crucial to improving the health and well-being of both mothers and their children.

A decade ago, promising data from the Manitoba study in Canada demonstrated the positive influence of cash allowances on improving maternal health during pregnancy and perinatal conditions. However, questions remain regarding whether these findings can be replicated in a post-pandemic U.S. context. In particular, there is limited understanding of the optimal timing and duration of prenatal stipend programs to maximize their impact on birth outcomes and child health during the first two years of life. While existing research sheds light on the benefits of financial support during pregnancy-such as improvements in birth outcomes, child immunization, and health behaviors in the first year-less is known about the long-term effects of cash allowances extending beyond delivery into the child's early years. Investigating this specific timeframe could provide valuable insights to inform policies aimed at reducing poverty and improving health outcomes for vulnerable populations.

This clinical trial seeks to explore the effects of providing direct financial support (unconditional cash transfers) to pregnant women on their health and the health of their babies. Specifically, the study will examine the impact of cash allowances on maternal physical and mental health, healthcare access, nutrition, and the child's growth and overall health during the first two years of life.

Participants will be randomly assigned to either a high cash or low cash group. Each participant will: (1) Complete a baseline survey upon enrollment (2) Complete a follow-up survey 12 months after enrollment. (3) Complete a final survey 18 months after enrollment.

Additionally, the study will review participants' medical records and may include qualitative interviews with some participants to better understand their experiences with cash support and health outcomes.

This research is conducted in collaboration with The Bridge Project (TBP), a New York-based non-governmental organization (NGO) founded in 2021, which offers unconditional cash transfers to mothers of infants born into poverty. This study will assess how these transfers impact maternal and child health outcomes. The findings of this study will provide critical data on the potential benefits of unconditional cash transfers for maternal and child health. These findings could inform public health policy and programs designed to alleviate poverty and promote health equity for vulnerable populations.

The researchers aim to:

* Evaluate the impact of a cash allowance program, initiated in the first trimester or second of pregnancy, on birth outcomes and toddler health.
* Assess the influence of cash allowances on maternal physical and mental health across the pre- and postnatal periods.
* Investigate the combined effects of cash allowances and health insurance on healthcare access and service utilization.
* Explore the role of cash allowances in improving the nutritional quality of diets among pregnant and breastfeeding mothers.

ELIGIBILITY:
Inclusion criteria for treatment and control

* Living in any of the study sites: Appalachian regions (West Virginia, Ohio, Kentucky, Tennessee)
* Being in the first or second trimester
* Being 18 years or older

Exclusion criteria

* Mothers with severe conditions such as terminal cancer.
* Mothers with identified addiction disorders. This includes any current or past addiction to legal (pain medication, alcohol) or illegal substance that has known risk for self-harm death (suicide, overdose) and/or consequences for maternal and/or fetal health.
* Mothers younger than 18 years old.
* Not living in the study site range
* Mothers incarcerated during the course of the study
* Mothers institutionalized during the course of the study.

Additional Notes:

* Participants who are not eligible for this study are also excluded from enrolling in the Bridge Project and receiving the direct cash transfer.
* Per protocol, participation in the study will be determined based on the inclusion and exclusion criteria. Final eligibility and study participation decisions will be made at the discretion of the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Preterm Babies | Immediately after birth
  Preterm birth is defined as a birth that occurs before 37 completed weeks of gestation. This outcome will assess the number of preterm births within the study population as documented in medical records.
Number of babies with low birth weight | Immediately after birth
  Low birth weight is defined as an infant born weighing less than 2,500 grams (approximately 5.5 pounds) at birth. This measure will assess the number of infants in the study who meet this criteria, as low birth weight is associated with increased risks of health complications for the newborn, such as developmental delays, respiratory issues, and long-term health challenges. Weight collected at time of birth as documented in medical records.
Score on Edinburgh Postnatal Depression Scale (EPDS) - Mothers Mental Health | Baseline, 12 months, 18 months
  The EPDS is a 10-item self-reported questionnaire designed to screen for symptoms of postnatal depression. Scores range from 0 to 30, with higher scores indicating greater depressive symptoms.
Number of Babies Admitted to the NICU | Immediately after birth
  This outcome will assess the number of infants requiring admission to the Neonatal Intensive Care Unit (NICU) after birth. Collected at birth, based on the number of babies admitted to the NICU as documented in medical records.
Gestational Age | Immediately after birth
  The mean gestational ages of the infants will be calculated. Gestational age refers to the length of time a baby has been in the womb, typically measured in weeks from the first day of the mother's last menstrual period (LMP) to the date of delivery. Gestational age will be collected at birth as documented in medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Monk, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
The intent is to create a repository. The Columbia repository protocol has not yet been created.